CLINICAL TRIAL: NCT05579496
Title: Rebooting Infant Pain Assessment: Using Machine Learning to Exponentially Improve Neonatal Intensive Care Unit Practice
Acronym: BabyAI
Status: Recruiting | Type: Observational
Sponsor: York University (Other)
Collaborators: MOUNT SINAI HOSPITAL (Other); University College, London (Other); University College London Hospitals (Other); University of Calgary (Other); McMaster University (Other)
Responsible Party: Principal Investigator, RRiddell, Full Professor, York University
Other Study IDs: 19-0252-A
Record Dates: First submitted 2020-12-24; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Acute Pain
Keywords: NICU (Neonatal Intensive Care Unit); Artificial Intelligence; Pain Assessment
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants Hospitalized in the NICU: Infants born between 28 0/7 weeks 32 6/7 weeks gestational age, who are within 6 weeks postnatal age, and their caregiver and/or health professional will be recruited for qualitative interview.

SUMMARY:
A multi-national multidisciplinary team will be working collaboratively to build a machine learning algorithm to distinguish between preterm infant distress states in the Neonatal Intensive Care Unit.

DETAILED DESCRIPTION:
Unmanaged pain in hospitalized infants has serious long-term complications. Our international team of knowledge users and health/natural science/engineering/social science researchers have come together to build a machine learning algorithm that will learn how to discriminate invasive and non-invasive distress. A sample of 400 preterm infants (300 from Mount Sinai Hospital and 100 from University College London Hospital [UCLH]) and their mothers will be followed during a routine painful procedure (heel lance). Pain indicators (facial grimacing [behavioural indicators], heart rate, oxygen saturation levels [physiologic indicators], brain electrical activity) during the painful procedure will be used to train the algorithm to discriminate between different types of distress (pain-related and non-pain related).

ELIGIBILITY:
* QUALITATIVE INTERVIEWS
* Inclusion Criteria:
* parents of a child currently in the NICU or
* health professionals currently working in the NICU.
* Exclusion Criteria:
* Participants who cannot communicate fluently in English
* QUANTITITATIVE DATA CAPTURE (video, eeg, ecg, SPo2)
* Inclusion Criteria:
* Infants born between 28 0/7 weeks 32 6/7 weeks gestational age
* Infants who are within 6 weeks postnatal age
* Infants who are undergoing a routine heel lance
* Exclusion Criteria:
* Infants with congenital malformations
* Infants receiving analgesics or sedatives at the time of study (aside from sucrose),
* Infants with history of perinatal hypoxia/ischemia at the time of study.
* Infants with diaper rash or excoriated buttocks

Ages: 27 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Behavioural Correlate of Distress | NFCS-P coded in 1-5 minute epochs, over 2 hour surrounding painful procedure (time locked to heel lance; approximately 1 hour before to 1 hour after heel lance)
  To be analyzed using machine learning via bedside videography: Facial Grimacing using Neonatal Facial Coding System(NFCS-P subset; Bucsea et al., in preparation)
Cortical Correlate of Distress | For 2 hours surrounding Painful procedure (time locked to heel lance; approximately 1 hour before to 1 hour after heel lance)
  To be analyzed using machine learning via bedside monitoring: Continuous EEG data capture
Cardiac Correlates of Distress | Over 2 hours surrounding Painful procedure (time locked to heel lance)
  To be analyzed using machine learning via bedside monitoring: Heart Rate, Heart Rate Variability
Oxygen Saturation Correlate of Distress | Over 2 hours surrounding Painful procedure (time locked to heel lance; approximately 1 hour before to 1 hour after heel lance)
  To be analyzed using machine learning via bedside monitoring: amount of oxygen-carrying hemoglobin in the blood relative to the amount of hemoglobin not carrying oxygen

SECONDARY OUTCOMES:
Semi-Structured Interview | These interviews are occurring at the beginning of the study and will be qualitatively analyzed. They are not linked to infants whose data we are collecting primary outcomes.
  Health Professionals and Caregivers will be asked about their thoughts on using AI for infant pain assessment

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Pillai Riddell, PhD, Principal Investigator — York University/Mount Sinai Hospital
Locations (2):
- Mount Sinai Hospital, Toronto, Ontario, Canada
- University College London Hospital, London, No Province, United Kingdom

IPD SHARING:
Plan to Share IPD: No